CLINICAL TRIAL: NCT06804031
Title: Nutrition and Exercise Education Given to Middle School Students on Adolescents' Health Literacy, Physical Activity and Healthy Eating Self-efficacy Levels: A Randomized Controlled Trial
Brief Title: Adolescents' Health Literacy, Physical Activity and Healthy Eating Self-efficacy Levels
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adem SÜMEN (Other)
Collaborators: Ministry of National Education, Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Adem SÜMEN, Associate Professor, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TBAEK-591
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obesity Prevention; Exercise; Nutrition; Health Literacy; Physical Activity; Self-Efficacy
Keywords: adolesence; nutrition; exercise; health literacy; physical activity; healthy eating; self-efficacy
MeSH Terms: conditions — Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (Experimental)
  Interventions: Behavioral: Nutrition and exercise education
- Control group (No Intervention)
- Control group 2 (No Intervention): At the end of the research, the data of control group I and control group II will be compared to evaluate whether there is an interaction.

INTERVENTIONS:
Behavioral: Nutrition and exercise education — Nutrition and exercise training was created as a result of literature review, and expert opinions (Public Health Nursing, Pediatric Nursing, Physical Therapy and Rehabilitation, Nutrition and Dietetics) were taken for the training content and finalized. The training program consists of six sessions. It is planned to have one session per week and each session will last 30-45 minutes on average. The times when the students are available will be determined by discussing with the school administration in advance. Computers and barcovisions in schools will be utilized for the training of students. Trainings will be conducted through verbal expression, power point presentations, brainstorming, exercises, games, written and visual materials, video screenings and question-answer methods. Adolescents will be given bookmarks, magnets and brochures prepared to prevent obesity.
  Arms: Experimental group

SUMMARY:
Adolescence is a critical transitional period characterized by rapid and multifaceted changes in physical, psychological, and social dimensions. According to the World Health Organization, adolescence encompasses the age range of 10 to 19 years. Alongside physical changes, this period involves significant developments and transformations in knowledge, skills, and behaviors, driven by the individual's identity formation process. Health behaviors such as nutrition and physical activity play a pivotal role in protecting and promoting adolescent health. However, unhealthy eating habits and insufficient physical activity are highly prevalent among adolescents.

These behaviors are associated with physical problems, including obesity, diabetes, hypertension, cardiovascular diseases, delayed growth and development, and psychological issues such as susceptibility to stress, low self-esteem, and lack of confidence. Consequently, fostering healthy eating and physical activity behaviors in adolescents is essential.

Given that adolescents spend a considerable portion of their time in school, implementing school-based interventions to promote these behaviors represents an effective approach to preventing lifestyle-related health issues in adulthood. The literature indicates that various interventions aimed at improving nutrition and physical activity behaviors in adolescents are generally effective. Nevertheless, sustaining these behaviors in the long term remains a challenge, as studies have shown that increases in knowledge do not always translate into behavioral changes.

One of the most effective strategies for instilling healthy behaviors in adolescents is health education. School-based health education not only facilitates the acquisition of functional health literacy but also strengthens the attitudes, beliefs, and practical skills necessary for adopting and maintaining healthy behaviors. Moreover, health education is a powerful tool for enhancing health literacy components such as accessing, understanding, evaluating, and utilizing accurate health information, enabling adolescents to take responsibility for their health and make informed decisions.

This study aims to contribute to fostering healthy eating and physical activity behaviors in adolescents, supporting their transformation into lifelong habits. Additionally, the findings are expected to guide school health professionals, particularly school nurses, in expanding interventions within the scope of school health services.

ELIGIBILITY:
Inclusion Criteria:

* - Volunteering to participate in the research
* Being allowed to participate in the study by their parents
* No physical or mental disabilities and chronic diseases (diabetes, metabolic syndrome, heart disease, etc.)

Exclusion Criteria:

* - Incomplete completion of research data collection forms
* Declining to participate in the research
* Failure to complete at least 5 health education sessions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Health Literacy Scale for School-Age Children | 5-6 month
  The health literacy scale for school-age children was developed to assess the health literacy of school-age children. The scale consists of 10 items and one dimension. The total score is between 10 and 40. The total score obtained from the scale (10-25 points) defines low health literacy, (26-35 points) medium health literacy, (36-40 points) high health literacy.
Physical Activity Self-Efficacy Scale for Children | 5-6 month
  It will be used to measure physical activity self-efficacy. The scale consists of 9 items. The score that can be obtained from the scale varies between 9-27, and the higher the score, the lower the strength of physical activity self-efficacy.
Healthy Eating Self-Efficacy Scale for Children | 5-6 month
  It was studied to be used in the assessment of children's self-efficacy for healthy eating. The scale consists of 9 items and one dimension. Participants can score between 0 and 18 points on the scale. The higher the scale score, the higher the self-efficacy for healthy eating.

SECONDARY OUTCOMES:
Adolescent Health Promotion Scale - Nutrition and Exercise Subscale | 5-6 month
  The scale was developed to assess the level of health promotion behavior of adolescents. The total score that can be obtained from the scale varies between 6-30 for the nutrition sub-dimension and between 4-20 for the exercise sub-dimension. A high total score in the nutrition subscale indicates that adolescents have positive nutrition behaviors, and a high total score in the exercise subscale indicates that adolescents have positive exercise behaviors.
Nutrition-Exercise Attitude Scale | 5-6 month
  The nutrition-exercise attitude scale was developed to evaluate the nutrition-exercise attitudes of adolescents. The total score that can be obtained from the scale varies between 13 and 65. A high total score indicates a positive attitude towards nutrition-exercise, while a low score indicates negative attitudes towards nutrition-exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz Universty, Kumluca, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No